CLINICAL TRIAL: NCT01249131
Title: A Phase I, Single-Dose, Randomized, Cross-Over, Relative Bioavailability, and Food Effect Study of GDC-0973 in Healthy Subjects
Brief Title: A Study of Relative Bioavailability and Food Effect Study of Cobimetinib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MEK4953g
Record Dates: First submitted 2010-11-24; First posted 2010-11-29 (Estimated); Results first posted 2016-07-18 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — cobimetinib

ARMS (6):
- Treatment A first, then Treatment B, followed by Treatment C (Experimental): Treatment A: One 20-mg tablet of cobimetinib will be administered orally with 240 milliliter (mL) room temperature water after at least an 8-hour fast, in first intervention period. Treatment B: Four 5-mg capsules of cobimetinib will be administered orally with 240 mL room temperature water after at least an 8-hour fast, in second intervention period. Treatment C: One 20-mg tablet of cobimetinib will be administered orally with 240 mL room temperature water within 30 minutes of eating a standard Food and Drug Administration (FDA) high-fat meal, in third intervention period. The washout period between each period will be a minimum of 10 days.
  Interventions: Drug: Cobimetinib
- Treatment A first, then Treatment C, followed by Treatment B (Experimental): Treatment A: One 20-mg tablet of cobimetinib will be administered orally with 240 mL room temperature water after at least an 8-hour fast, in first intervention period. Treatment C: One 20-mg tablet of cobimetinib will be administered orally with 240 mL room temperature water within 30 minutes of eating a standard FDA high-fat meal, in second intervention period. Treatment B: Four 5-mg capsules of cobimetinib administered will be orally with 240 mL room temperature water after at least an 8-hour fast, in third intervention period.
  Interventions: Drug: Cobimetinib
- Treatment B first, then Treatment A, followed by Treatment C (Experimental): Treatment B: Four 5-mg capsules of cobimetinib will be administered orally with 240 mL room temperature water after at least an 8-hour fast, in first intervention period. Treatment A: One 20-mg tablet of cobimetinib will be administered orally with 240 mL room temperature water after at least an 8-hour fast, in second intervention period. Treatment C: One 20-mg tablet of cobimetinib will be administered orally with 240 mL room temperature water within 30 minutes of eating a standard FDA high-fat meal, in third intervention period.
  Interventions: Drug: Cobimetinib
- Treatment B first, then Treatment C, followed by Treatment A (Experimental): Treatment B: Four 5-mg capsules of cobimetinib will be administered orally with 240 mL room temperature water after at least an 8-hour fast, in first intervention period. Treatment C: One 20-mg tablet of cobimetinib will be administered orally with 240 mL room temperature water within 30 minutes of eating a standard FDA high-fat meal, in second intervention period. Treatment A: One 20-mg tablet of cobimetinib will be administered orally with 240 mL room temperature water after at least an 8-hour fast, in third intervention period.
  Interventions: Drug: Cobimetinib
- Treatment C first, then Treatment A, followed by Treatment B (Experimental): Treatment C: One 20-mg tablet of cobimetinib will be administered orally with 240 mL room temperature water within 30 minutes of eating a standard FDA high-fat meal, in first intervention period. Treatment A: One 20-mg tablet of cobimetinib will be administered orally with 240 mL room temperature water after at least an 8-hour fast, in second intervention period. Treatment B: Four 5-mg capsules of cobimetinib will be administered orally with 240 mL room temperature water after at least an 8-hour fast, in third intervention period.
  Interventions: Drug: Cobimetinib
- Treatment C first, then Treatment B, followed by Treatment A (Experimental): Treatment C: One 20-mg tablet of cobimetinib will be administered orally with 240 mL room temperature water within 30 minutes of eating a standard FDA high-fat meal, in first intervention period. Treatment B: Four 5-mg capsules of cobimetinib will be administered orally with 240 mL room temperature water after at least an 8-hour fast, in second intervention period. Treatment A: One 20-mg tablet of cobimetinib will be administered orally with 240 mL room temperature water after at least an 8-hour fast, in third intervention period.
  Interventions: Drug: Cobimetinib

INTERVENTIONS:
Drug: Cobimetinib — Cobimetinib 20 mg will be given orally as tablet formulation in fasted or fed state, or as capsule formulation in fasted state.
  Other Names: GDC-0973; XL518

SUMMARY:
This study will be an open-label, randomized, 3-way, 6-sequence crossover study in healthy participants for determining the relative bioavailability of the tablet formulation to the capsule formulation and the effect of food on the relative bioavailability of the tablet formulation.

ELIGIBILITY:
Inclusion Criteria

* Within body mass index range 18.5 to 29.9 kilograms per meter square (kg/m^2)
* In good health, determined by no clinically significant findings from medical history, 12-lead electrocardiogram (ECG) and vital signs
* Clinical laboratory evaluations within the reference range for the test laboratory
* Negative test for selected drugs of abuse at Screening and at each Check-in
* Negative hepatitis panel and anti-hepatitis C virus and negative human immunodeficiency virus (HIV) antibody screens
* Healthy males and females of non-child-bearing potential or who agree to use effective contraception

Exclusion Criteria

* Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs except that appendectomy, hernia repair, and cholecystectomy will be allowed
* History or presence of an abnormal ECG
* History of alcoholism or drug addiction prior to study start
* Use of any tobacco-containing or nicotine-containing products prior to study start
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 28 days or 5 half-lives, whichever is longer, prior to study start
* Use of any prescription medications/products, including proton pump inhibitors, within 14 days prior to study start
* Poor peripheral venous access
* Any acute or chronic condition that would limit the participant's ability to complete and/or participate in this clinical study
* Female participant is pregnant, lactating, or breastfeeding
* Predisposing factors to retinal vein occlusion (RVO)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2011-01-10 (Actual); Study Completion 2011-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Rooney, M.D., PhD, Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A First, Then Treatment B, Followed by Treatment C: Treatment A: One 20-milligram (mg) tablet of cobimetinib administered orally with 240 milliliter (mL) room temperature water after at least an 8-hour fast, in first intervention period. Treatment B: Four 5-mg capsules of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast, in second intervention period. Treatment C: One 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water within 30 minutes of eating a standard Food and Drug Administration (FDA) high-fat meal, in third intervention period. The washout period between each period was a minimum of 10 days.
- Treatment A First, Then Treatment C, Followed by Treatment B: Treatment A: One 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast, in first intervention period. Treatment C: One 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water within 30 minutes of eating a standard FDA high-fat meal, in second intervention period. Treatment B: Four 5-mg capsules of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast, in third intervention period.
- Treatment B First, Then Treatment A, Followed by Treatment C: Treatment B first, then Treatment A, followed by Treatment C Treatment B: Four 5-mg capsules of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast, in first intervention period. Treatment A: One 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast, in second intervention period. Treatment C: One 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water within 30 minutes of eating a standard FDA high-fat meal, in third intervention period.
- Treatment B First, Then Treatment C, Followed by Treatment A: Treatment B first, then Treatment C, followed by Treatment A Treatment B: Four 5-mg capsules of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast, in first intervention period. Treatment C: One 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water within 30 minutes of eating a standard FDA high-fat meal, in second intervention period. Treatment A: One 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast, in third intervention period.
- Treatment C First, Then Treatment A, Followed by Treatment B: Treatment C: One 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water within 30 minutes of eating a standard FDA high-fat meal, in first intervention period. Treatment A: One 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast, in second intervention period. Treatment B: Four 5-mg capsules of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast, in third intervention period.
- Treatment C First, Then Treatment B, Followed by Treatment A: Treatment C: One 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water within 30 minutes of eating a standard FDA high-fat meal, in first intervention period. Treatment B: Four 5-mg capsules of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast, in second intervention period. Treatment A: One 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast, in third intervention period.
Period: First Intervention
Arm/Group | Treatment A First, Then Treatment B, Followed by Treatment C | Treatment A First, Then Treatment C, Followed by Treatment B | Treatment B First, Then Treatment A, Followed by Treatment C | Treatment B First, Then Treatment C, Followed by Treatment A | Treatment C First, Then Treatment A, Followed by Treatment B | Treatment C First, Then Treatment B, Followed by Treatment A
Started | 3 | 3 | 4 | 3 | 3 | 4
Completed | 3 | 3 | 4 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period of 10 Days
Arm/Group | Treatment A First, Then Treatment B, Followed by Treatment C | Treatment A First, Then Treatment C, Followed by Treatment B | Treatment B First, Then Treatment A, Followed by Treatment C | Treatment B First, Then Treatment C, Followed by Treatment A | Treatment C First, Then Treatment A, Followed by Treatment B | Treatment C First, Then Treatment B, Followed by Treatment A
Started | 3 | 3 | 4 | 3 | 3 | 4
Completed | 3 | 3 | 4 | 3 | 2 | 4
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Period: Second Intervention
Arm/Group | Treatment A First, Then Treatment B, Followed by Treatment C | Treatment A First, Then Treatment C, Followed by Treatment B | Treatment B First, Then Treatment A, Followed by Treatment C | Treatment B First, Then Treatment C, Followed by Treatment A | Treatment C First, Then Treatment A, Followed by Treatment B | Treatment C First, Then Treatment B, Followed by Treatment A
Started | 3 | 3 | 4 | 3 | 2 | 4
Completed | 3 | 3 | 4 | 3 | 2 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period of 10 Days
Arm/Group | Treatment A First, Then Treatment B, Followed by Treatment C | Treatment A First, Then Treatment C, Followed by Treatment B | Treatment B First, Then Treatment A, Followed by Treatment C | Treatment B First, Then Treatment C, Followed by Treatment A | Treatment C First, Then Treatment A, Followed by Treatment B | Treatment C First, Then Treatment B, Followed by Treatment A
Started | 3 | 3 | 4 | 3 | 2 | 4
Completed | 3 | 3 | 4 | 3 | 2 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Treatment A First, Then Treatment B, Followed by Treatment C | Treatment A First, Then Treatment C, Followed by Treatment B | Treatment B First, Then Treatment A, Followed by Treatment C | Treatment B First, Then Treatment C, Followed by Treatment A | Treatment C First, Then Treatment A, Followed by Treatment B | Treatment C First, Then Treatment B, Followed by Treatment A
Started | 3 | 3 | 4 | 3 | 2 | 4
Completed | 3 | 3 | 4 | 3 | 2 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Entire Study Population: All participants randomized to any treatment.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 36 [19 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf)
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - inf). It is obtained from AUC (0 - t) plus AUC (t - inf).
Time Frame: Day 1 at 0 hour (predose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 hours postdose
Population: Pharmacokinetic parameters populations included all enrolled participants. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (ng*hr/mL)
Groups:
- Cobimetinib One 20 mg Tablet [Fasted]: One 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast.
- Cobimetinib Four 5 mg Capsules [Fasted]: Four 5-mg capsules of cobimetinib administered orally with 240 mL room temperature water after at least an 8-hour fast.
- Cobimetinib One 20 mg Tablet [Fed]: One 20-mg tablet of cobimetinib administered orally with 240 mL room temperature water within 30 minutes of eating a standard FDA high-fat meal.
Arm/Group | Cobimetinib One 20 mg Tablet [Fasted] | Cobimetinib Four 5 mg Capsules [Fasted] | Cobimetinib One 20 mg Tablet [Fed]
Number analyzed (Participants) | 19 | 18 | 20
nanograms*hours/milliliter (ng*hr/mL) | 780 (34.7) | 717 (45.1) | 858 (42.4)
Statistical Analysis 1: Comparison: Cobimetinib One 20 mg Tablet [Fasted] vs Cobimetinib Four 5 mg Capsules [Fasted]; Test type: Superiority or Other; Ratio of Least Squares (LS) Means (in %) = 94.7, 90% CI 2-sided [83.9 to 107] — LS mean was calculated from analysis of variance (ANOVA). Data for dose-normalized AUCinf were natural log-transformed prior to analysis. Ratio of AUCinf LS means for log-transformed parameter (expressed as a percent)
Statistical Analysis 2: Comparison: Cobimetinib One 20 mg Tablet [Fasted] vs Cobimetinib One 20 mg Tablet [Fed]; Test type: Superiority or Other; Ratio of LS Means (in %) = 110, 90% CI 2-sided [98.2 to 124] — LS mean was calculated from ANOVA. Data for dose-normalized AUCinf were natural log-transformed prior to analysis. Ratio of AUCinf LS means for log-transformed parameter (expressed as a percent)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Day 1 at 0 hour (predose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Cobimetinib One 20 mg Tablet [Fasted] | Cobimetinib Four 5 mg Capsules [Fasted] | Cobimetinib One 20 mg Tablet [Fed]
Number analyzed (Participants) | 19 | 18 | 20
nanograms per milliliter (ng/mL) | 16.0 (33.5) | 14.9 (45.9) | 17.2 (43.1)
Statistical Analysis 1: Comparison: Cobimetinib One 20 mg Tablet [Fasted] vs Cobimetinib Four 5 mg Capsules [Fasted]; Test type: Superiority or Other; Ratio of LS Means (in %) = 96.9, 90% CI 2-sided [84.2 to 111] — LS mean was calculated from ANOVA. Data for dose-normalized Cmax were natural log-transformed prior to analysis. Ratio of Cmax LS means for log-transformed parameter (expressed as a percent)
Statistical Analysis 2: Comparison: Cobimetinib One 20 mg Tablet [Fasted] vs Cobimetinib One 20 mg Tablet [Fed]; Test type: Superiority or Other; Ratio of LS Means (in %) = 107, 90% CI 2-sided [93.8 to 123] — [estimate comment as in outcome 2, analysis 1]

3. Primary Outcome: Minimum Observed Plasma Concentration (Cmin)
Time Frame: Day 1 at 0 hour (predose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cobimetinib One 20 mg Tablet [Fasted] | Cobimetinib Four 5 mg Capsules [Fasted] | Cobimetinib One 20 mg Tablet [Fed]
Number analyzed (Participants) | 5 | 7 | 5
ng/mL | 0.307 (46.6) | 0.36 (56.6) | 0.361 (60.3)

4. Primary Outcome: Apparent Oral Clearance (CL/F)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Day 1 at 0 hour (predose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour (L/hr)
Arm/Group | Cobimetinib One 20 mg Tablet [Fasted] | Cobimetinib Four 5 mg Capsules [Fasted] | Cobimetinib One 20 mg Tablet [Fed]
Number analyzed (Participants) | 19 | 18 | 20
Liters per hour (L/hr) | 25.6 (34.7) | 25.2 (45.1) | 23.3 (42.4)

5. Primary Outcome: Apparent Volume of Distribution (V/F)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Day 1 at 0 hour (predose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Cobimetinib One 20 mg Tablet [Fasted] | Cobimetinib Four 5 mg Capsules [Fasted] | Cobimetinib One 20 mg Tablet [Fed]
Number analyzed (Participants) | 19 | 18 | 20
Liters (L) | 2103 (40.4) | 1930 (50.2) | 1900 (38.3)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from start of study treatment in first period to end of last period (up to 30 days)
Description: One participant discontinued study in first period and did not receive Cobimetinib One 20 mg Tablet [Fasted] in second period and Cobimetinib Four 5 mg Capsules [Fasted] in third period. Therefore, only 19 participants were evaluable for adverse events in these treatment arms.
Arm/Group | Cobimetinib One 20 mg Tablet [Fasted] | Cobimetinib Four 5 mg Capsules [Fasted] | Cobimetinib One 20 mg Tablet [Fed]
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 6/19 | 9/19 | 8/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cobimetinib One 20 mg Tablet [Fasted] (N=19) | Cobimetinib Four 5 mg Capsules [Fasted] (N=19) | Cobimetinib One 20 mg Tablet [Fed] (N=20)
Nausea (Gastrointestinal disorders) | 1 | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1
Vitreous detachment (Eye disorders) | 0 | 0 | 1
Chills (General disorders) | 1 | 1 | 0
Vessel puncture site haematoma (General disorders) | 1 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1
Vessel puncture site pain (General disorders) | 1 | 0 | 0
Vessel puncture site reaction (General disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.